CLINICAL TRIAL: NCT05318092
Title: Evaluating the Safety and Efficacy of the AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE for Treatment of Acute Pulmonary Embolism
Acronym: APEX-AV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-EVT-01
Record Dates: First submitted 2022-03-24; First posted 2022-04-08 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Embolism; Acute Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE (Experimental): Single Arm Study - Use of AngioDynamics' AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE for the treatment of acute pulmonary embolism
  Interventions: Device: AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE

INTERVENTIONS:
Device: AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE — The AngioDynamics' AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE has five main components, a flexible cannula (F1885), sheath, tapered obturator, aspirator handle, and waste bag.

SUMMARY:
To evaluate the safety and effectiveness of percutaneous mechanical aspiration thrombectomy using the AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE in a prospective trial of patients with acute intermediate-risk pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form.
* 18 years of age and older.
* Clinical signs and symptoms consistent with acute intermediate-risk pulmonary embolism for less than or equal to 14 days.
* Diagnosis of pulmonary embolism detected from computed tomography angiography (CTA).
* Right Ventricle to Left Ventricle (RV/LV) ratio of 0.9 or higher.
* Systolic blood pressure (SBP) of 90 mmHg or higher
* Heart rate of 130 beats per minute (BPM) or less prior to the procedure.
* Deemed medically eligible for interventional procedure(s) per institutional guidelines and/or clinical judgment.

Exclusion Criteria:

Excluded from the study if he/she meets any of the following exclusion criteria

* May be pregnant as determined by a positive pregnancy test or who are breastfeeding.
* Has any contraindication to systemic or therapeutic doses of heparin or anticoagulants.
* Has used thrombolytics (tPA) in the past 30 days of baseline CTA.
* Has pulmonary hypertension with peak pulmonary artery pressure (PAP) > 70 mmHg.
* Fraction of inspired oxygen (FiO2) requirement >40% or >6 liters per minute (LPM) to keep oxygen saturations >90%
* Hematocrit <28% within 6 hours of the index procedure.
* Platelets count < 100,000/µL.
* Serum creatinine >1.8 mg/dL.
* International Normalized Ratio (INR) > 3
* Has undergone a major trauma within the past 14 days of the index procedure and have Injury Severity Score (ISS) > 15.
* Presence of cancer requiring active chemotherapy.
* Known bleeding diathesis or coagulation disorder.
* Has had a cardiovascular or pulmonary surgery within the past 7 days of index procedure.
* History of severe or chronic pulmonary hypertension, uncompensated heart failure, chest irradiation, underlying lung disease that is oxygen dependent, Heparin-induced thrombocytopenia (HIT) and/or chronic left heart disease with left ventricular ejection fraction ≤ 30%.
* Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated.
* Requires Vasopressor after fluids to keep pressure ≥ 90 mmHg.
* With left bundle branch block.
* Has intracardiac lead in the right ventricle or atrium.
* Evidence such as imaging or other that suggests the subject is not appropriate for this procedure.
* Has life expectancy < 90 days.
* Dependent on extracorporeal life support such as extracorporeal membrane oxygenation (ECMO).
* Participation in another investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - HonorHealth, Scottsdale, Arizona
  - UCLA Health, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - HCA Memorial Hospital Jacksonville, Jacksonville, Florida
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - OSF Healthcare, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Oshner Medical Center, Jefferson, Louisiana
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Rutgers University, Newark, New Jersey
  - University of Buffalo, Buffalo, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Kettering Health, Miamisburg, Ohio
  - UPMC Hamot, Erie, Pennsylvania
  - Einstein Medical Center, Montgomery, Pennsylvania
  - UPMC Pittsburgh, Pittsburgh, Pennsylvania
  - Tennova Healthcare -Turkey Creek Medical Center, Knoxville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Memorial Hermann (University of Texas at Houston), Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Aurora Health Care, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System: AngioDynamics' AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Period: Overall Study
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Started | 122
Completed | 118
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: As Treated Population - all subjects who met the inclusion/exclusion criteria of the study and in whom the AlphaVac MMA F1885 cannula was placed within the jugular or one of the common femoral veins.
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 84
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 122
Baseline Right Ventricle to Left Ventricle (RV/LV) Ratio [Mean (Standard Deviation); unit: ratio] — Core lab-adjudicated baseline Right Ventricle to Left Ventricle (RV/LV) ratio
  ratio | 1.5 (0.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Ventricle to Left Ventricle (RV/LV) Ratio Between Baseline and 48 Hours Post-procedure Assessed by Computed Tomography Angiography (CTA)
Description: Change in Right Ventricle to Left Ventricle (RV/LV) ratio between baseline and 48 hours post-procedure assessed by Computed Tomography Angiography (CTA) and read by the study's core lab.
Time Frame: At 48 hours post-procedure
Population: Modified As Treated population - all subjects who met the inclusion/exclusion criteria of the study and in whom the AlphaVac MMA F1885 cannula was placed within the jugular or one of the common femoral veins, who did not receive thrombolytics during the index procedure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 119
ratio | -0.45 (0.27)

2. Primary Outcome: Rate of Major Adverse Events (MAEs) Within 48 Hours After the Index Procedure.
Description: Rate of Major Adverse Events (MAEs) within the first 48 hours after the index procedure, defined as:
  Device-related death Major bleeding
  Device-related SAEs of:
  * Clinical Deterioration
  * Pulmonary Vascular Injury
  * Cardiac Injury
Time Frame: Within 48 hours post-procedure
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 122
Participants
  Subjects experiencing a MAE | 5
  Subjects not experiencing a MAE | 117

3. Secondary Outcome: Use of Thrombolytics Within 48 Hours of the Procedure.
Description: Use of thrombolytics within 48 hours of the procedure.
Time Frame: Within 48 hours of the procedure
Population: Modified As Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 119
Participants | 0

4. Secondary Outcome: Length of Stay in the Intensive Care Unit (ICU)/Hospital Within 30 Days Post-procedure.
Description: Length of stay in the Intensive care unit (ICU)/Hospital within 30 days post-procedure.
Time Frame: Within 30 days of the procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 119
days
  Length of Stay in ICU | 1.4 (1.7)
  Length of Stay in Hospital | 5.2 (3.3)

5. Secondary Outcome: Change in Modified Miller Index Between Baseline and 48 Hours Post-procedure Assessed by Computed Tomography Angiography (CTA).
Description: Change in Modified Miller Index between baseline and 48 hours post-procedure assessed by Computed Tomography Angiography (CTA) and read by the study's core lab. Modified Miller Index ranges from 0 - 16 (higher values mean higher thrombus burden) and a greater negative change is a better outcome.
Time Frame: At 48 hours post-procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 119
score on a scale | -5.6 (4.3)

6. Secondary Outcome: Rate of Device Related Complications Including Clinical Deterioration, Cardiac Injury, Pulmonary Vascular Injury, Major Bleeding, and Device-related Death Within 48 Hours of the Index Procedure.
Description: Rate of device related complications including clinical deterioration, cardiac injury, pulmonary vascular injury, major bleeding, and device-related death within 48 hours of the index procedure.
Time Frame: Within 48 hours of the procedure
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 122
Participants
  Device-related clinical deterioration: Subjects with event | 1
  Device-related clinical deterioration: Subjects without event | 121
  Device-related pulmonary vascular injury: Subjects with event | 1
  Device-related pulmonary vascular injury: Subjects without event | 121
  Device-related cardiac injury: Subjects with event | 1
  Device-related cardiac injury: Subjects without event | 121
  Major bleeding: Subjects with event | 5
  Major bleeding: Subjects without event | 117
  Device-related death: Subjects with event | 0
  Device-related death: Subjects without event | 122

7. Secondary Outcome: Rate of Device-related Serious Adverse Events (SAEs) and Death for Any Cause Within 30 Days Post-procedure.
Description: Rate of device-related Serious Adverse Events (SAEs) and death for any cause within 30 days post-procedure.
Time Frame: Within 30 days of the procedure
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 122
Participants
  Device-related SAEs: Subjects with event | 4
  Device-related SAEs: Subjects without event | 118
  Death for any cause: Subjects with event | 0
  Death for any cause: Subjects without event | 122

8. Secondary Outcome: Symptomatic Pulmonary Embolism (PE) Recurrence Within 30 Days.
Description: Symptomatic PE recurrence within 30 days.
Time Frame: Within 30 days of the procedure
Population: As Treated population - all subjects who met the inclusion/exclusion criteria of the study and in whom the AlphaVac MMA F1885 cannula was placed within the jugular or one of the common femoral veins - who completed the study through 30 days (n=118).
Measure: Count of Participants; unit: Participants
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Number analyzed (Participants) | 118
Participants | 1

ADVERSE EVENTS:
Time Frame: 30 days (+/- 7 days) post-procedure
Arm/Group | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 18/122
Other Adverse Events (participants affected / at risk) | 9/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System (N=122)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcus test positive (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 5 (5)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System (N=122)
Deep vein thrombosis (Vascular disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of the results from any single site experience within the study is not allowed until the preparation and publication of the multi-center results. Exceptions to this rule require the prior written approval of the Sponsor. If after 180 days from the conclusion of the study, the Sponsor has not published the results, the investigators may publish without prior approval from the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT05318092/Prot_SAP_000.pdf